CLINICAL TRIAL: NCT02804945
Title: A Pilot Study of Mesenchymal Stem Cells for Treatment of Acute Respiratory Distress Syndrome in Patients With Malignancies
Brief Title: Mesenchymal Stem Cells (MSCs) for Treatment of Acute Respiratory Distress Syndrome (ARD) in Patients With Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Katz Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0327; NCI-2016-01184 (Other: NCI CTRP)
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Blood And Marrow Transplantation; Adult Respiratory Distress Syndrome
Keywords: Blood And Marrow Transplantation; Adult Respiratory Distress Syndrome; ARDS; Allogeneic human mesenchymal stem cells; hMSCs; Placebo; Plasma-Lyte A solution; Standard of Care; Recent onset pulmonary toxicity
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stem Cells (Experimental): Participants receive Mesenchymal Stem Cells (MSCs) for adult respiratory distress syndrome (ARDS).
  Participants receive a maximum dose of 3 x 10^6 cell/Kg by vein one time on Day 1.
  Interventions: Biological: Mesenchymal Stem Cells (MSCs)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSCs) — Participants receive a maximum dose of 3 x 10^6 cell/Kg by vein one time on Day 1.

SUMMARY:
The goal of this clinical research study is to learn about the safety of giving mesenchymal stem cells (MSCs) to patients who have ARDS. Researchers also want to learn if these cells can help control ARDS when given with drugs that are routinely used to treat ARDS.

In this study, participants will receive 1 infusion of MSCs.

This is an investigational study. MSC infusions for the treatment of ARDS is investigational.

Up to 20 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
The MSCs:

MSCs are a type of stem cell that can be removed from bone marrow and grown into many different cell types that can be used to treat cancer and other diseases. The MSCs used in this study were collected from healthy donors and are stored and grown in a laboratory at MD Anderson. The product you will receive is from a healthy donor that is not related to you.

MSC Administration:

If you are found to be eligible to take part in this study, you will receive MSCs by vein over about 1-2 hours 1 time on Day 1.

Study Visits:

On Days 1 and 3:

* Blood (about 2 tablespoons) will be drawn for routine tests, to check your heart, kidney, and liver function, and for biomarker testing.
* Blood (about ½ teaspoon) will be drawn to check the oxygen level in your blood.

On Days 14 and 30:

°Blood (about 2 tablespoons) will be drawn for routine tests, to check your heart, kidney, and liver function, and for biomarker testing.

On Days 30 and 60:

°You will be checked for possible reactions to your treatment, including graft-versus-host disease (GVHD - a reaction of the donor's immune cells against your body). This will be checked by physical exam, by the doctor reviewing your side effects, and blood from standard of care blood draws.

Length of Study:

Your participation on this study will end after the Day 60 study visit. You will be taken off study early if you are not able to receive the MSC infusion(s), if intolerable side effects occur, if the doctor thinks it is in your best interest, or if you are unable to follow study directions.

ELIGIBILITY:
Inclusion Criteria:

1. ARDS characterized by hypoxemia and bilateral radiographic opacities not fully explained by cardiac failure or fluid overload as judged by the treating physician using all available data. Moderate ARDS includes patients with malignancies with the previous presentation and a P/F ratio </= 200 or SF ratio of </= 214. The duration of the hypoxemia criterion and the radiograph criterion must be within 10 days of the time of enrollment.
2. Patients age >/=18 years.
3. Treated with appropriate maximal medical therapy for pulmonary toxicity.
4. Negative pregnancy test in a woman with childbearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
5. Patient or legally appropriate proxy must be able to understand study instructions and sign consent.

Exclusion Criteria:

1. Unstable ventricular tachycardia or fibrillation.
2. Moribund patients not expected to survive up to 48 hours.
3. Patients with ARDS resulting from trauma.
4. Patients with documented deep venous thrombosis or pulmonary embolism within the past 3 months.
5. Patients with severe chronic liver disease (Childs-Pugh score > 10).
6. Patients with previous solid organ transplant.
7. Pregnant and/or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Adverse Events of Participants Treated with Allogeneic Human Mesenchymal Stem Cells (hMSCs) With Acute Respiratory Distress Syndrome (ARD) | 30 days
  Adverse Events determined by CTCAE version 4.

SECONDARY OUTCOMES:
Clinical Improvement of Participants Treated with Allogeneic Human Mesenchymal Stem Cells (hMSCs) With Acute Respiratory Distress Syndrome (ARD) | Baseline, 7 days and 30 days
  Clinical improvement defined as decreased mechanical ventilation after the mesenchymal stem cell (MSC) infusion.
Improvement in PF or S/F Ratio of Participants Treated with Allogeneic Human Mesenchymal Stem Cells (hMSCs) With Acute Respiratory Distress Syndrome (ARD) | Baseline, 7 days and 30 days
  An improvement in PF or S/F ratio defined as decreased mechanical ventilatory requirement.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L. Olson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org